CLINICAL TRIAL: NCT00515034
Title: A Randomized, Open-Label, Multicenter Study to Assess the Safety and Tolerability of Doripenem Compared With Imipenem in the Treatment of Subjects With Complicated Intra-Abdominal Infections or Ventilator Associated Pneumonia
Brief Title: A Safety and Tolerability Study of Doripenem in Patients With Abdominal Infections or Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Senior Director Clinical Development, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012934; DORINOS2001
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2011-05

CONDITIONS: Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Pneumonia; Abdominal Abscess; Bacterial Infections
Keywords: Doripenem; Imipenem; Cilastatin; Vancomycin; DORIBAX, DORIPREX, FINIBAX, DURAPTA, PRIMAXIN, Anti Bacterial Agents; Ileus; Hospitalized; Fever
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Pneumonia; Abdominal Abscess; Bacterial Infections; Ileus; Fever | interventions — Cilastatin, Imipenem Drug Combination; Doripenem

ARMS (4):
- 001 (Experimental): Doripenem 1 gram infused over 4 hours at 8-hour intervals for patients with Ventilator-Associated Pneumonia (VAP) for 7 to 14 days Vancomycin and/or amikacin may be added as adjunctive therapy as per investigator discretion
  Interventions: Drug: Doripenem
- 002 (Active Comparator): Imipenem/cilastatin 1 gram infused over 1 hour at 8 hour intervals for patients with Ventilator-Associated Pneumonia (VAP) for 7 to 14 days Vancomycin and/or amikacin may be added as adjunctive therapy as per investigator discretion
  Interventions: Drug: Imipenem/cilastatin
- 003 (Experimental): Doripenem 1 gram infused over 4 hours at 8 hour intervals for patients with complicated intrabdominal infections (cIAI) for 5 to 14 days Vancomycin may be added as adjunctive therapy as per investigator discretion
  Interventions: Drug: Doripenem
- 004 (Active Comparator): Imipenem/cilastatin 1 gram infused over 1 hour at 8 hour intervals for patients with complicated intrabdominal infections (cIAI) for 5 to 14 days Vancomycin may be added as adjunctive therapy as per investigator discretion
  Interventions: Drug: Imipenem/cilastatin

INTERVENTIONS:
Drug: Imipenem/cilastatin — Vancomycin and/or amikacin may be added as adjunctive therapy as per investigator discretion
  Arms: 002
Drug: Imipenem/cilastatin — Vancomycin and/or amikacin may be added as adjunctive therapy as per investigator discretion
  Arms: 004
Drug: Doripenem — 1 gram infused over 4 hours at 8-hour intervals for patients with Ventilator-Associated Pneumonia (VAP) for 7 to 14 days
  Arms: 001
Drug: Doripenem — 1 gram infused over 1 hour at 8 hour intervals for patients with Ventilator-Associated Pneumonia (VAP) for 7 to 14 days
  Arms: 003

SUMMARY:
The purpose of this study is to assess the safety and tolerability of doripenem compared to imipenem in Ventilator-assisted pneumonia and complicated Intra-abdominal Infection. The study population will include hospitalized patients (or patients resident in a chronic health care facility) who have a diagnosis of either Ventilator associated pneumonia or complicated Intra-abdominal Infection.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all people involved know the identity of the intervention), multicenter study that will evaluate the safety and tolerability of doripenem (an antibiotic used to treat infections) in patients with ventilator-associated pneumonia (VAP) or complicated intra-abdominal infection (cIAI). Approximately 250 patients will be assigned in a 3:1 ratio to receive doripenem or imipenem/cilastatin (188 patients randomized to receive doripenem and 62 patients randomized to receive imipenem/cilastatin). Furthermore, patients who receive doripenem or imipenem/cilastatin will be stratified by disease (VAP or cIAI). Therefore, for reporting purposes, there will be 4 groups: Patients with VAP treated with doripenem, patients with VAP treated with imipenem/cilastatin, patients with cIAI treated with doripenem, and patients with cIAI treated with imipenem/cilastatin. Study drug will be administered intravenously (iv) (through a vein) for 7 to 14 days for patients with VAP and for 5 to 14 days for patients with cIAI. The maximum duration of study drug is 14 days. Vancomycin and/or amikacin may be added to the study drug regimen as adjunctive therapy for those patients who meet study specified criteria. The recommended dosage of vancomycin is 1 g every 12 hours administered by iv infusion. The addition of amikacin is at the discretion of the investigator for patients with VAP (not cIAI) and the recommended dosing regimen for amikacin is 15 mg/kg given iv once a day. Alternative amikacin regimens or other aminoglycoside regimens may be permitted. Safety will be assessed during the study by the monitoring of adverse events, evaluation of laboratory test results, and changes in vital signs. The primary endpoint of this study is to assess the overall incidence of treatment-emergent adverse events (TEAEs) from the initiation of the first infusion of study drug and up to 30 days after the completion of study drug therapy. Treatment-emergent adverse events are defined as adverse events that occur or worsen between the initial infusion of study drug up to 30 days after the last dose of study drug. The hypothesis for this study is that doripenem has a similar safety profile to imipenem. Doripenem (1g at 8-hour intervals over a period of 4 hours) or imipenem/cilastatin (1g at 8-hours over a period of 1 hour) will be administered by intravenous (iv) infusion (delivery of drug slowly into the vein over a period of time). Patients diagnosed with ventilator associated pneumonia (VAP) will be treated for 7 to 14 days and patients with complicated intra-abdominal infections (cIAI) will be treated for 5 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be hospitalized with a diagnosis of Ventilator-Assisted Pneumonia (VAP) or complicated Intra-Abdominal Infection (cIAI)
* Patients with VAP must have been hospitalized (or been in a chronic care facility) for >= 5 days, have received mechanical ventilation for >= 48 hours, have a Clinical Pulmonary Infection Score (CPIS) of >= 5, have new or progressive radiographic infiltrates (not related to another disease process)
* Patients with cIAI must have clinical evidence of intra-abdominal infection, abdominal pain or tenderness, localized or diffuse abdominal wall rigidity, mass, ileus or have a requirement for surgical intervention (e.g., laparotomy, laparoscopic surgery, or percutaneous draining of an abscess) within 24 hours of study entry

Exclusion Criteria:

* Patients with a history of acute hepatic failure or acute decompensation of chronic hepatic failure, history of severe impairment of renal function, history of immunocompromising illness, acquired immunodeficiency syndrome (AIDS), or human immunodeficiency virus (HIV) with a CD4 count less than 200 cells/mL within the past 6 months
* organ (including bone marrow) transplant recipients
* hematologic malignancy
* use of immunosuppressive therapy at screening, including use of high dose corticosteroids (e.g., > 40 mg prednisone or equivalent per day for > 2 weeks)
* history of any rapidly progressing disease or immediately life-threatening illness (including acute hepatic failure and septic shock)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Groups:
- VAP Treated With Doripenem: Doripenem 1 g infused over 4 hours at 8-hour intervals for patients with Ventilator-Associated Pneumonia (VAP) for 7-14 days
- VAP Treated With Imipenem/Cilastatin: Imipenem/cilastatin 1 g infused over 1 hour at 8-hour intervals for patients with Ventilator-Associated Pneumonia (VAP)for 7-14 days
- cIAI Treated With Doripenem: Doripenem 1 g infused over 4 hours at 8-hour intervals for patients with complicated Intra-Abdominal Infection (cIAI) for 5-14 days
- cIAI Treated With Imipenem/Cilastatin: Imipenem/cilastatin 1 g infused over 1 hour at 8-hour intervals for patients with complicated Intra-Abdominal Infection (cIAI) for 5-14 days
Period: Overall Study
Arm/Group | VAP Treated With Doripenem | VAP Treated With Imipenem/Cilastatin | cIAI Treated With Doripenem | cIAI Treated With Imipenem/Cilastatin
Started | 49 | 15 | 62 | 20
TREATED | 48 | 15 | 61 | 19
Completed | 41 | 13 | 54 | 15
Not Completed | 8 | 2 | 8 | 5
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Death | 4 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAP Treated With Doripenem | VAP Treated With Imipenem/Cilastatin | cIAI Treated With Doripenem | cIAI Treated With Imipenem/Cilastatin | Total
Number analyzed (Participants) | 49 | 15 | 62 | 20 | 146
Age, Customized [Number; unit: participants]
  <65 years | 35 | 11 | 48 | 16 | 110
  >=65 years | 14 | 4 | 14 | 4 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 25 | 5 | 48
  Male | 37 | 9 | 37 | 15 | 98
Region of Enrollment [Number; unit: participants]
  North America | 14 | 3 | 24 | 7 | 48
  Europe | 19 | 7 | 15 | 4 | 45
  South America | 16 | 5 | 23 | 9 | 53

OUTCOME MEASURES:

1. Primary Outcome: Patients With Incidence of Treatment-emergent Adverse Events (TEAEs).
Description: Treatment-emergent adverse events (TEAEs) are defined as AEs with onset dates on or after the date of the start of the infusion of first dose of study therapy and within 30 days after administration of the last dose of study therapy.
Time Frame: from the initiation of the first infusion of study drug therapy and up to 30 days after the completion of study drug therapy
Population: population is the as-treated analysis set - that is subjects who were administered therapy
Measure: Number; unit: participants
Arm/Group | VAP Treated With Doripenem | VAP Treated With Imipenem/Cilastatin | cIAI Treated With Doripenem | cIAI Treated With Imipenem/Cilastatin
Number analyzed (Participants) | 48 | 15 | 61 | 19
participants | 42 | 13 | 37 | 15

2. Secondary Outcome: Patients With VAP Who Were Clinically Cured
Description: clinical cure is the complete resolution of signs and symptoms of pneumonia or lack of progression of chest x-ray abnormalities to such an extent that no further antimicrobial therapy was necessary.
Time Frame: 7 to 14 days after the end of IV therapy
Population: the population is the number of participants who are clinically evaluable
Measure: Number; unit: participants
Arm/Group | VAP Treated With Doripenem | VAP Treated With Imipenem/Cilastatin | cIAI Treated With Doripenem | cIAI Treated With Imipenem/Cilastatin
Number analyzed (Participants) | 25 | 9 | 0 | 0
participants | 16 | 7 |  |
Statistical Analysis 1: Comparison: VAP Treated With Doripenem vs VAP Treated With Imipenem/Cilastatin; There is no formal hypothesis test for this outcome. Only summary data are provided; Test type: Non-Inferiority or Equivalence — Percent of participants who are clinically cured including 95% confidence intervals are provided; normal approximation to the binomial; Risk Difference (RD) = -13.8, 95% CI 2-sided [-54.4 to 26.8] — Treatment difference (doripenem minus imipenem/cilastatin) in percent of participants who are clinically cured

3. Secondary Outcome: Patients With cIAI Who Were Clinically Cured
Description: clinical cure is the complete resolution or significant improvement of signs or symptoms of cIAI, such that no additional antimicrobial therapy or surgical or percutaneous intervention is required for the treatment of the current infection.
Time Frame: 7 to 14 days after the end of IV therapy
Population: participants who were clinically evaluable
Measure: Number; unit: participants
Arm/Group | VAP Treated With Doripenem | VAP Treated With Imipenem/Cilastatin | cIAI Treated With Doripenem | cIAI Treated With Imipenem/Cilastatin
Number analyzed (Participants) | 0 | 0 | 47 | 14
participants |  |  | 39 | 9
Statistical Analysis 1: Comparison: cIAI Treated With Doripenem vs cIAI Treated With Imipenem/Cilastatin; There is no formal hypothesis test for this outcome. Only summary data are presented; Test type: Non-Inferiority or Equivalence — Percent of participants who are clinically cured including 95% confidence intervals are provided; normal approximation to binomial; Risk Difference (RD) = 18.7, 95% CI 2-sided [-13.2 to 50.6] — Treatment difference (doripenem minus imipenem) in percent of participants who are clinically cured

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated informed consent form was obtained until 30 days after the completion of study drug therapy
Arm/Group | VAP Treated With Doripenem | VAP Treated With Imipenem/Cilastatin | cIAI Treated With Doripenem | cIAI Treated With Imipenem/Cilastatin
Serious Adverse Events (participants affected / at risk) | 16/48 | 4/15 | 11/61 | 7/19
Other Adverse Events (participants affected / at risk) | 42/48 | 13/15 | 37/61 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAP Treated With Doripenem (N=48) | VAP Treated With Imipenem/Cilastatin (N=15) | cIAI Treated With Doripenem (N=61) | cIAI Treated With Imipenem/Cilastatin (N=19)
Autonomic Nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
bradyarrhythmia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
colonic fistura (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gasrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypoglycaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAP Treated With Doripenem (N=48) | VAP Treated With Imipenem/Cilastatin (N=15) | cIAI Treated With Doripenem (N=61) | cIAI Treated With Imipenem/Cilastatin (N=19)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 1 (1) | 1 (1) | 1 (1)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 3 (3) | 1 (1)
hypertension (Vascular disorders) | 2 (2) | 1 (1) | 7 (7) | 2 (2)
hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 4 (4) | 3 (3)
hypotension (Vascular disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (6) | 0 (0)
pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
pyrexia (General disorders) | 5 (5) | 2 (2) | 5 (5) | 3 (3)
urinary tract infection (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Viomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Oedema Peripheral (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Urinary Tract Infection Fungal (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
open-label study design and limited number of subjects in the comparator group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days